CLINICAL TRIAL: NCT03745586
Title: Giant Cell Arteritis Treatment With Ultra-short Glucocorticoids and Tocilizumab
Acronym: GUSTO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00845
Record Dates: First submitted 2018-11-06; First posted 2018-11-19 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — tocilizumab; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All study participants (Experimental)
  Interventions: Drug: Tocilizumab; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Tocilizumab — Day 3: Tocilizumab infusion (8mg/kg body-weight) Day 10- week 52: Tocilizumab s.c. injections (162mg) in weekly intervals
Drug: Glucocorticoids — Day0-day2: methylprednisolone 500mg i.v.

SUMMARY:
Two recent RCTs showed the ability of tocilizumab to induce and maintain remission of giant cell arteritis. Both studies used the dosing schemes for Rheumatoid Arthritis (i.e. 8mg/kg bodyweight i.v. in 4-weekly intervals and 162mg weekly s.c., respectively). In both trials glucocorticoids (GC) were initially administrated at medium to high doses with subsequent rapid reduction and discontinuation over 24 weeks. In case of relapse, GC doses were re-increased.

The results of both studies suggest that GC could be reduced more rapidly. This would further reduce GC-induced adverse effects.

Thus, the investigators propose to perform an open label single arm study to assess the efficacy of ultra-short co-medication with GC, using Simon's minimax two-stage design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly onset Giant Cell Arteritis (GCA) with diagnosis of GCA within 4 weeks before screening visit, satisfying ACR criteria and a CRP > 25 mg/L AND biopsy proven GCA (according to ACR criteria) OR a large vessel vasculitis assessed by MR Angiography (MRA) or PET/CT (PET).
2. Previous treatment with GC for a maximum of 10 days since diagnosis of GCA at a maximal dose of 60 mg/day of prednisone or equivalent.
3. Patient's written informed consent.

Exclusion Criteria:

1. Rheumatic diseases (except for CPPD/chondrocalcinosis) other than GCA or polymyalgia rheumatica (i.e., RA, autoimmune connectivitides, other systemic vasculitides, a.o.)
2. Chronic use of systemic CS with inability, in the opinion of the investigator, to withdraw CS treatment at day 4 according to protocol
3. Evidence of significant and/or uncontrolled concomitant disease such as, but not limited to, cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine (in particular diabetes mellitus) or gastrointestinal disorders (including previous complicated diverticulitis) which, in the investigator's opinion, would preclude patient participation or impact the benefit-risk ratio
4. Any condition or general state of health which, in the Investigator's opinion, would preclude participation in the study
5. Actual or recent myocardial infarction (within the last 3 months before screening visit)
6. Significant cardiac disease (NYHA Class III and IV), known severe chronic obstructive pulmonary disease (COPD) (FEV1 < 50% predicted or Functional dyspnea > Grade 3 on the MRC Dyspnea Scale) or other significant pulmonary disease
7. Uncontrolled disease (such as asthma, psoriasis or inflammatory bowel disease) where flares are commonly treated with oral or injectable corticosteroids
8. Known active infection of any kind, or any major episode of infection requiring hospitalization or treatment with i.v. anti-infectives within 4 weeks of baseline or completion of oral anti-infectives within 2 weeks before screening visit
9. History of deep space/tissue infection (e.g. fasciitis, abscess, osteomyelitis) within 52 weeks before screening visit
10. Any surgical procedure, including bone/joint surgery within 8 weeks prior before screening visit or planned within the duration of the study
11. History of serious recurrent or chronic infection (for screening for a chest infection a chest radiograph will be performed at screening if not performed within 12 weeks before screening visit
12. Lack of peripheral venous access
13. Body weight > 150 kg or BMI > 35
14. Previous treatment with tocilizumab or any other biological agent within last 6 months before screening visit; Rituximab within 12 months before screening visit
15. Treatment with any investigational agent within 28 days of screening visit or 5 half-lives of the investigational drug (whichever is the longer)
16. History of severe allergic or anaphylactic reaction to any biologic agent or known hypersensitivity to any component of tocilizumab
17. Receipt of any vaccine within 28 days prior to screening visit (a patient's vaccination record and need for immunization prior to receiving tocilizumab/placebo must be carefully investigated)
18. Positive tests for hepatitis B surface antigen (HBsAg) or hepatitis C serology
19. Positive Quantiferon-TB test for latent Tb without subsequent INH prophylaxis
20. Patients with active Tb which had to be treated for Tb within 2 years before the screening visit
21. Absolute neutrophil count (ANC) < 2.0 x 103/L, white blood cells < 2.5 x 103/L, platelet count < 100,000/L
22. Hemoglobin < 8.0 g/dL
23. Concentrations of serum IgG and/or IgM below 5.0 mg/mL and 0.40 mg/mL, respectively
24. Serum creatinine > 2.0 mg/dL
25. Alanine aminotransferase (ALT) or aspartate amino-transferase (AST) > 1.5 times the upper limit of normal (ULN)
26. Total bilirubin > 1.5 times the upper limit of normal (ULN)
27. Triglycerides > 400 mmol/dL (non-fasted) or > 250 mmol/dL (fasted) at screening
28. Premenopausal status and nursing (definition of postmenopausal status: Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child-bearing potential)
29. Technical implants such as cardiac pacemakers (for MR-angiogram)
30. Claustrophobia (for MR-angiogram)
31. Known allergy against the contrast media (Multihance® or Dotarem® as alternative)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Remission | Week 24
  Proportion of patients achieving remission within 31 days and without relapse until week 24

SECONDARY OUTCOMES:
Remission | Week 24 and week 52
  Proportion of patients with complete relapse-free remission of disease at week 24 and at week 52
Time to first relapse | through study completion, an average of 1 year
  Time to first relapse

CONTACTS AND LOCATIONS:
Overall Officials: Peter Villiger, Prof, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christ L, Seitz L, Scholz G, Sarbu AC, Amsler J, Butikofer L, Tappeiner C, Kollert F, Reichenbach S, Villiger PM. Tocilizumab monotherapy after ultra-short glucocorticoid administration in giant cell arteritis: a single-arm, open-label, proof-of-concept study. Lancet Rheumatol. 2021 Sep;3(9):e619-e626. doi: 10.1016/S2665-9913(21)00152-1. Epub 2021 Jul 2. PMID 38287611
- [Derived] Christ L, Gloor AD, Kollert F, Gaber T, Buttgereit F, Reichenbach S, Villiger PM. Serum proteomics in giant cell arteritis in response to a three-day pulse of glucocorticoid followed by tocilizumab monotherapy (the GUSTO trial). Front Immunol. 2023 May 23;14:1165758. doi: 10.3389/fimmu.2023.1165758. eCollection 2023. PMID 37287970
- [Derived] Seitz L, Christ L, Lotscher F, Scholz G, Sarbu AC, Butikofer L, Kollert F, Schmidt WA, Reichenbach S, Villiger PM. Quantitative ultrasound to monitor the vascular response to tocilizumab in giant cell arteritis. Rheumatology (Oxford). 2021 Nov 3;60(11):5052-5059. doi: 10.1093/rheumatology/keab484. PMID 34117737